CLINICAL TRIAL: NCT00177424
Title: Intervention to Prevent Post-Stroke Major Depression.
Brief Title: Sertraline for Preventing Post-stroke Depression and Improving Rehabilitation Outcomes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment goals could not be met.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K23MH067710-02 (NIH); K23MH067710-02 (NIH); 0310068; DATR AK-TNGP1
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2009-02

CONDITIONS: Cerebrovascular Accident; Depression
Keywords: Rehabilitation
MeSH Terms: conditions — Stroke; Depression | interventions — Sertraline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Sertraline
  Interventions: Drug: sertraline
- 2 (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sertraline — Subjects will initially be started on either sertraline 12.5mg/d or placebo and will receive this dose for 3 days. Subjects will then be increased to 25mg/d for 4 days, then 50mg/d for 7 days, then increased to 75mg/d. Seventy-five mg per day is the target dose for the remainder of the subject's participation in the study. The study medication will not be titrated past 75mg/d.
  Arms: 1
Drug: Placebo — matching placebo tablets
  Arms: 2

SUMMARY:
This study will determine the effectiveness of sertraline administration after a stroke in preventing the onset of post-stroke depression.

DETAILED DESCRIPTION:
Persons who suffer from a stroke are at high risk for developing post-stroke major depression (PSMD), an illness that has a negative impact on post-stroke physical rehabilitation and is associated with increased morbidity and mortality. Unfortunately, early detection and successful treatment of post-stroke major depression improves, but does not normalize, stroke rehabilitation outcomes compared to stroke survivors who never developed post-stroke depression. Therefore, preventing the onset of PSMD and its associated disability is an attractive possibility. This study is a placebo controlled, 10-month double-blind trial of sertraline in the prevention of PSMD in stroke survivors, with a 2-month naturalistic continuation phase. The primary outcome will be the incidence of Major Depression post-stroke. Additional outcomes will include the severity of depressive symptoms post-stroke and the level of disability experienced by the two treatment groups. An exploratory analysis will also be conducted to elucidate participant characteristics that may be moderators of the participants' response to the preventive intervention, thereby refining the profile of disabled stroke survivors most likely to benefit from the preventive intervention.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00781326

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke within 3 months of study entry
* Admitted to a UPMC hospital for acute inpatient treatment or rehabilitation of stroke
* Speaks English
* Females willing to use an effective form of birth control throughout the study

Exclusion Criteria:

* Meets DSM-IV-TR criteria for a major depressive episode
* History of any bipolar disorder
* Psychotic or history of a psychotic disorder
* Meets DMS-IV TR criteria for alcohol or substance abuse or dependence criteria within 3 months of study entry
* Current treatment with antidepressant medication for any reason (e.g., anxiety disorder, neuropathic pain)
* Primary hemorrhagic stroke
* Language impairment severe enough to prevent valid neuropsychiatric assessment
* History of another CNS disease other than prior stroke or psychiatric illness (e.g., head trauma, multiple sclerosis, HIV with CNS involvement)
* Pulse <50 or >100 beats per minute
* Significant hyponatremia (Na <130meq)
* Current hypothyroid state
* Medically unstable including symptoms of delirium (determined by review of the subject's medical status with the treating (clinical) physician; standard blood chemistry lab work will be obtained if not checked within the preceding 30 days)
* History of sensitivity to sertraline
* Pregnant or breastfeeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the incidence of Major Depression post-stroke. | 12 months

SECONDARY OUTCOMES:
Additional outcomes will include the severity of depressive symptoms post-stroke as measured by the Hamilton Depression Rating Scale, and the level of disability experienced by the two treatment groups, as measured by the Functional Independence Measure. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ellen M Whyte, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: The American Stroke Association website provides general information to stroke survivors and their families. — http://www.strokeassociation.org